CLINICAL TRIAL: NCT00950989
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-dose Study to Evaluate the Safety, Tolerability, and Efficacy of AMG 827 in Subjects With Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Brief Title: Brodalumab (AMG 827) in Rheumatoid Arthritis (RA) Participants With Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20090061
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Autoimmune Diseases; Musculoskeletal Diseases; Joint Diseases; Arthritis; Connective Tissue Diseases; Arthritis, Rheumatoid; Rheumatic Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases; Musculoskeletal Diseases; Joint Diseases; Arthritis; Connective Tissue Diseases; Rheumatic Diseases | interventions — brodalumab; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Placebo on day 1 and weeks 1, 2, 4, 6, 8, and 10 for a total of 7 doses plus a stable weekly dose of methotrexate and folic acid supplementation (at least 5 mg per week).
  Interventions: Drug: Placebo; Drug: Methotrexate; Dietary Supplement: folic acid
- Brodalumab 70 mg (Experimental): 70 mg brodalumab on day 1 and weeks 1, 2, 4, 6, 8, and 10 for a total of 7 doses plus a stable weekly dose of methotrexate and folic acid supplementation (at least 5 mg per week).
  Interventions: Drug: Brodalumab; Drug: Methotrexate; Dietary Supplement: folic acid
- Brodalumab 140 mg (Experimental): 140 mg brodalumab on day 1 and weeks 1, 2, 4, 6, 8, and 10 for a total of 7 doses plus a stable weekly dose of methotrexateand folic acid supplementation (at least 5 mg per week).
  Interventions: Drug: Brodalumab; Drug: Methotrexate; Dietary Supplement: folic acid
- Brodalumab 210 mg (Placebo Comparator): 210 mg brodalumab on day 1 and weeks 1, 2, 4, 6, 8, and 10 for a total of 7 doses plus a stable weekly dose of methotrexate and folic acid supplementation (at least 5 mg per week).
  Interventions: Drug: Brodalumab; Drug: Methotrexate; Dietary Supplement: folic acid

INTERVENTIONS:
Drug: Brodalumab — 3 single subcutaneous (SC) injections at day 1 and weeks 1, 2, 4, 6, 8, and 10
  Other Names: AMG 827
  Arms: Brodalumab 140 mg; Brodalumab 210 mg; Brodalumab 70 mg
Drug: Placebo — 3 single SC injections at day 1 and weeks 1, 2, 4, 6, 8, and 10
  Arms: Placebo
Drug: Methotrexate — Two methotrexate dose adjustments were allowed in the event of methotrexate toxicity, however, doses < 7.5 mg/week necessitated discontinuation from study.
Dietary Supplement: folic acid — at least 5 mg per week

SUMMARY:
Study in participants with RA who have an inadequate response to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Active RA for least 6 months
* Current RA defined as ≥ 6 swollen joints (out of 66 joints examined) and ≥ 8 tender/painful joints (out of 68 joints examined) at screening and baseline (swollen and tender/painful joint count must not include distal interphalangeal joints) and at least 1 of the following at screening: Erythrocyte sedimentation rate ≥ 28 mm or C-reactive protein > 15 mg/L
* At least 1 of the following at screening: Rheumatoid factor positive or Anti-cyclic citrullinated peptide antibody positive
* Currently taking methotrexate for ≥ 12 weeks and on a stable dose of methotrexate at 15 to 25 mg weekly for ≥ 4 weeks at day -1.

Exclusion Criteria:

* Prosthetic joint infection within 5 years of screening or native joint infection within 1 year of screening
* Class IV RA
* Felty's syndrome
* Presence of serious infection
* Significant concurrent medical conditions
* Pregnant or breast feeding
* Significant Laboratory abnormalities
* Any disease-modifying anti-rheumatic drug (DMARD) other than methotrexate within 28 days
* Leflunomide or live vaccines within 3 months
* Previous use of any experimental or commercially available biologic DMARD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2009-12-30 (Actual); Primary Completion 2011-02-11 (Actual); Study Completion 2011-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Pavelka K, Chon Y, Newmark R, Lin SL, Baumgartner S, Erondu N. A study to evaluate the safety, tolerability, and efficacy of brodalumab in subjects with rheumatoid arthritis and an inadequate response to methotrexate. J Rheumatol. 2015 Jun;42(6):912-9. doi: 10.3899/jrheum.141271. Epub 2015 Apr 15. PMID 25877498
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the following countries: Bulgaria, Canada, Czech Republic, Hungary, Latvia, Mexico, Poland, United Kingdom, United States.
Pre-assignment Details: Participants were randomized in a 1:1:1:1 ratio to receive brodalumab (doses of 70, 140, or 210 mg) or placebo. Randomization was stratified by sex with enrollment of women limited to 200 participants.
Groups:
- Brodalumab 140 mg: 140 mg brodalumab on day 1 and weeks 1, 2, 4, 6, 8, and 10 for a total of 7 doses plus a stable weekly dose of methotrexate and folic acid supplementation (at least 5 mg per week).
Period: Overall Study
Arm/Group | Placebo | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Started | 63 | 63 | 63 | 63
Completed | 59 | 60 | 60 | 63
Not Completed | 4 | 3 | 3 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Administrative Decision | 0 | 1 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg | Total
Number analyzed (Participants) | 63 | 63 | 63 | 63 | 252
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 57 | 60 | 53 | 58 | 228
  >= 65 years | 6 | 3 | 10 | 5 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 50 | 49 | 50 | 200
  Male | 12 | 13 | 14 | 13 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 48 | 53 | 50 | 56 | 207
  Black or African American | 1 | 1 | 1 | 0 | 3
  Hispanic or Latino | 14 | 8 | 12 | 6 | 40
  Asian | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: A positive ACR50 response is defined if the following 3 criteria for improvement from baseline were met:
  * 50% improvement in 68 tender joint count;
  * 50% improvement in 66 swollen joint count; and
  * 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of joint pain (measured on a 100 mm visual analog scale [VAS]),
    * Patient's global assessment of disease activity (measured on a 0-10 Likert scale),
    * Physician's global assessment of disease activity (measured on a 0-10 Likert scale),
    * Patient's self assessment of disability (Health Assessment Questionnaire - Disability Index [HAQ-DI]),
    * Acute phase reactant: erythrocyte sedimentation rate (ESR) or C-Reactive Protein (CRP), whichever has bigger improvement.
Time Frame: Baseline, week 12
Population: Full Analysis Set: all randomized participants with an assessment. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Number analyzed (Participants) | 63 | 63 | 63 | 63
percentage of participants | 12.7 | 15.9 | 15.9 | 9.5
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 70 mg; Test type: Superiority; p = 0.598, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rate = 3.2, 95% CI 2-sided [-9.0 to 15.4]
Statistical Analysis 2: Comparison: Placebo vs Brodalumab 70 mg; Test type: Superiority; p = 0.993, Sequential testing + Hommel procedure — Adjusted p-value is based on a combination of sequential testing and the Hommel procedure to control the overall significance level for all the comparisons
Statistical Analysis 3: Comparison: Placebo vs Brodalumab 140 mg; Test type: Superiority; p = 0.635, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rate = 3.2, 95% CI 2-sided [-9.0 to 15.4]
Statistical Analysis 4: Comparison: Placebo vs Brodalumab 140 mg; Test type: Superiority; p = 0.740, Sequential testing + Hommel procedure — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.572, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rate = -3.2, 95% CI 2-sided [-14.1 to 7.8]
Statistical Analysis 6: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.572, Sequential testing + Hommel procedure — [p-value comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: A positive ACR20 response is defined if the following 3 criteria for improvement from baseline were met:
  * 20% improvement in 68 tender joint count;
  * 20% improvement in 66 swollen joint count; and
  * 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of joint pain (measured on a 100 mm visual analog scale [VAS]),
    * Patient's global assessment of disease activity (measured on a 0-10 Likert scale),
    * Physician's global assessment of disease activity (measured on a 0-10 Likert scale),
    * Patient's self assessment of disability (Health Assessment Questionnaire - Disability Index [HAQ-DI]),
    * Acute phase reactant: erythrocyte sedimentation rate (ESR) or C-Reactive Protein (CRP), whichever has bigger improvement.
Time Frame: Baseline, Week 12
Population: Full Analysis Set: all randomized participants with an assessment. Non-responder imputation.
Measure: Number; unit: percentage of partcipants
Arm/Group | Placebo | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Number analyzed (Participants) | 63 | 63 | 63 | 63
percentage of partcipants | 42.9 | 39.7 | 36.5 | 46.0
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 70 mg; Test type: Superiority; p = 0.728, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rates = -3.2, 95% CI 2-sided [-20.4 to 14.0]
Statistical Analysis 2: Comparison: Placebo vs Brodalumab 70 mg; Test type: Superiority; p = 0.993, Sequential testing + Hommel procedure — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Brodalumab 140 mg; Test type: Superiority; p = 0.412, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rates = -6.3, 95% CI 2-sided [-23.4 to 10.7]
Statistical Analysis 4: Comparison: Placebo vs Brodalumab 140 mg; Test type: Superiority; p = 0.740, Sequential testing + Hommel procedures — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.740, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rates = 3.2, 95% CI 2-sided [-14.2 to 20.5]
Statistical Analysis 6: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.993, Sequential testing + Hommel procedure — [p-value comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: A positive ACR70 response is defined if the following 3 criteria for improvement from baseline were met:
  * 70% improvement in 68 tender joint count;
  * 70% improvement in 66 swollen joint count; and
  * 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of joint pain (measured on a 100 mm visual analog scale [VAS]),
    * Patient's global assessment of disease activity (measured on a 0-10 Likert scale),
    * Physician's global assessment of disease activity (measured on a 0-10 Likert scale),
    * Patient's self assessment of disability (Health Assessment Questionnaire - Disability Index [HAQ-DI]),
    * Acute phase reactant: erythrocyte sedimentation rate (ESR) or C-Reactive Protein (CRP), whichever has bigger improvement.
Time Frame: Baseline, week 12
Population: Full Analysis Set: all randomized participants with an assessment. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Number analyzed (Participants) | 63 | 63 | 63 | 63
percentage of participants | 3.2 | 3.2 | 3.2 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 70 mg; Test type: Superiority; p = 0.984, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rates = 0.0, 95% CI 2-sided [-6.1 to 6.1]
Statistical Analysis 2: Comparison: Placebo vs Brodalumab 70 mg; Test type: Superiority; p = 0.993, Sequential testing + Hommel procedure — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Brodalumab 140 mg; Test type: Superiority; p = 0.993, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rates = 0.0, 95% CI 2-sided [-6.1 to 6.1]
Statistical Analysis 4: Comparison: Placebo vs Brodalumab 140 mg; Test type: Superiority; p = 0.993, Sequential testing + Hommel procedure — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.159, Cochran-Mantel-Haenszel — P-value is nominal p-value without multiplicity adjustment based on Cochran-Mantel-Haenszel test adjusting for sex; Difference in response rates = -3.2, 95% CI 2-sided [-7.5 to 1.2]
Statistical Analysis 6: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.797, Sequential testing + Hommel procedure — [p-value comment as in outcome 1, analysis 2]

4. Secondary Outcome: Disease Activity Score 28 (DAS28) at Week 12
Description: The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables: • The number of tender joints assessed using the 28-jount count and number of swollen joints assessed using the 28-joint count; • Erythrocyte sedimentation rate (ESR); • Patient's global assessment of disease activity (measured on a 0-10 Likert scale). The DAS28 score ranges from 0 to 10, with higher scores indicating more severe disease activity.
Time Frame: Week 12
Population: Full Analysis Set: all randomized participants with an assessment. Last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Number analyzed (Participants) | 63 | 61 | 63 | 63
score on a scale | 5.0 (0.2) | 4.9 (0.2) | 5.1 (0.2) | 5.1 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 70 mg; Test type: Superiority; p = 0.459, ANCOVA — P-value is nominal without multiplicity adjustment based on ANCOVA model adjusting for sex and baseline DAS28 score; LS Mean of difference = -0.2, 95% CI 2-sided [-0.7 to 0.3], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo vs Brodalumab 140 mg; Test type: Superiority; p = 0.906, ANCOVA — P-value is nominal without multiplicity adjustment based on ANCOVA model adjusting for sex and baseline DAS28 score; LS mean of difference = 0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.849, ANCOVA — P-value is nominal without multiplicity adjustment based on ANCOVA model adjusting for sex and baseline DAS28 score; LS mean of difference = 0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.2

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation
Description: AEs are defined as any untoward medical occurrence, that does not necessarily have a causal relationship with this treatment. SAEs are defined as an AE that: is fatal; is life threatening (places the subject at immediate risk of death); requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; other significant medical hazard. The severity of events were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v 4.0: mild=grade 1, moderate=grade 2, severe=grade 3, life-threatening=grade 4, death=grade 5.
Time Frame: From first dose of study drug until the end of study; median (min, max) duration was 113 days (8, 132).
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Number analyzed (Participants) | 63 | 63 | 63 | 63
Participants
  AEs | 32 | 32 | 40 | 32
  SAEs | 2 | 1 | 1 | 3
  Fatal AEs | 0 | 0 | 1 | 0
  AEs leading to Study Discontinuation | 2 | 1 | 2 | 0
  AEs leading to Study Drug Discontinuation | 1 | 1 | 1 | 2
  CTCAE Grades 3, 4, 5 AEs | 4 | 3 | 2 | 4
  AEs Related to Study Drug | 12 | 8 | 14 | 11
  SAEs Related to Study Drug | 0 | 0 | 0 | 0
  Fatal AEs Related to Study Drug | 0 | 0 | 0 | 0
  AEs Related to Study Drug Leading to Study Discontinuation | 1 | 1 | 0 | 0
  AEs Related to Study Drug Leading to Study Drug Discontinuation | 0 | 1 | 0 | 2
  CTCAE Grades 3, 4, 5 AEs Related to Study Drug | 0 | 1 | 0 | 0

6. Secondary Outcome: Pharmacokinetics (PK) of Brodalumab: Maximum Observed Concentration (Cmax)
Time Frame: Week 8: Day 59-Day 61 (44-100 hours post-dose), Day 64 (160-176 hours post-dose), Week 10: pre-dose
Population: Participants who received brodalumab with an evaluable PK measurement.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Number analyzed (Participants) | 15 | 13 | 12
µg/mL | 3.02 (1.61) | 7.85 (4.37) | 17.9 (12.8)

7. Secondary Outcome: PK of Brodalumab: Time to Maximum Observed Concentration (Tmax)
Time Frame: Week 8: Day 59-Day 61 (44-100 hours post-dose), Day 64 (160-176 hours post-dose), Week 10: pre-dose
Population: Participants who received brodalumab with an evaluable PK measurement.
Measure: Median (Full Range); unit: days
Arm/Group | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Number analyzed (Participants) | 15 | 13 | 12
days | 1.94 [1.84 to 3.73] | 2.00 [1.84 to 6.92] | 1.96 [1.91 to 6.99]

8. Secondary Outcome: PK of Brodalumab: Area Under the Curve During the Dosing Interval (AUCtau)
Time Frame: Week 8: Day 59-Day 61 (44-100 hours post-dose), Day 64 (160-176 hours post-dose), Week 10: pre-dose
Population: Participants who received AMG 827 with an evaluable PK measurement.
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Number analyzed (Participants) | 15 | 13 | 12
µg*day/mL | 18.1 (15.2) | 73.3 (52.7) | 199 (161)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until the end of study; median (min, max) duration was 113 days (8, 132).
Arm/Group | Placebo | Brodalumab 70 mg | Brodalumab 140 mg | Brodalumab 210 mg
Serious Adverse Events (participants affected / at risk) | 2/63 | 1/63 | 1/63 | 3/63
Other Adverse Events (participants affected / at risk) | 18/63 | 19/63 | 25/63 | 12/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Brodalumab 70 mg (N=63) | Brodalumab 140 mg (N=63) | Brodalumab 210 mg (N=63)
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Brodalumab 70 mg (N=63) | Brodalumab 140 mg (N=63) | Brodalumab 210 mg (N=63)
Injection site pain (General disorders) | 4 | 2 | 2 | 2
Nasopharyngitis (Infections and infestations) | 2 | 3 | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 5 | 3
Urinary tract infection (Infections and infestations) | 1 | 2 | 5 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5 | 4 | 7 | 0
Headache (Nervous system disorders) | 4 | 3 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 1
Hypertension (Vascular disorders) | 4 | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.